CLINICAL TRIAL: NCT01197378
Title: A Long-Term, Open-Label, Safety and Efficacy Study of Cysteamine Bitartrate Delayed-release Capsules (RP103) in Patients With Cystinosis
Brief Title: Long-Term Safety Follow-up Study of Cysteamine Bitartrate Delayed-release Capsules (RP103)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP103-04; 2010-018365-34 (EudraCT Number)
Record Dates: First submitted 2010-09-03; First posted 2010-09-09 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cystinosis
Keywords: cystinosis; cysteamine; inheritable disease; orphan disease; CTNS protein, human; metabolic disease; nephropathic cystinosis
MeSH Terms: conditions — Cystinosis; Rare Diseases; Metabolic Diseases | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cysteamine Bitartrate (Experimental): Cysteamine bitartrate delayed-release capsules were administered twice daily for up to 96 months.
  Interventions: Drug: Cysteamine Bitartrate Delayed-release Capsules

INTERVENTIONS:
Drug: Cysteamine Bitartrate Delayed-release Capsules — Participants who entered the trial from the RP103-03 study continued treatment with cysteamine bitartrate every 12 hours at the last dose level prescribed during their participation in that study.
  Participants not entering the trial from Study RP103-03 were started on twice a day administration of cysteamine bitartrate at a total daily RP103 dose of 70% of their pre-study total daily stable Cystagon® dose.
  Other Names: RP103; PROCYSBI®

SUMMARY:
Cystinosis is an inherited disease that if untreated, results in kidney failure as early as the first decade of life. The current marketed therapy is Cystagon® (cysteamine bitartrate immediate release) which must be taken every six hours for the rest of the patient's life to prevent complications of cystinosis. Cysteamine bitartrate delayed-release capsules (RP103) is a formulation of cysteamine bitartrate that is being studied to see if it can be given less frequently, once every 12 hours, and have similar results to four times a day Cystagon®.

DETAILED DESCRIPTION:
This is a long-term, open-label, study to determine the safety and tolerability of twice a day treatment with cysteamine bitartrate delayed-release capsules (RP103). It will involve 6-9 monthly clinic visits followed by quarterly clinic visits for the duration of the study and home use of cysteamine bitartrate delayed-release capsules.

Initially, enrollment was open to those patients who had completed the previous Phase 3 Study (RP103-03, NCT01000961). Subsequently enrollment in Study RP103-04 was opened to additional participants, including children aged 1 to 6 years and renal transplant recipients, who had previously been on a stable dose of Cystagon® for at least 21 days.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects must have completed the last visit of Study RP103-03 and be willing to continue with RP103 treatment.

OR for patients who did not complete the RP103-03 study:

* Male and female subjects must have cystinosis.
* Subjects must be on a stable dose of Cystagon® at least 21 days prior to Screening.
* Within the last 6 months, no clinically significant change from normal in liver function tests (i.e., alanine aminotransferase [ALT], aspartate aminotransferase [AST], total bilirubin) and renal function (i.e., estimated glomerular filtration rate [eGFR]) at Screening as determined by the Investigator.
* Subjects with an eGFR corrected for body surface area > 30 mL/min/1.73m².
* Sexually active female subjects of childbearing potential (i.e., not surgically sterile [tubal ligation, hysterectomy, or bilateral oophorectomy] or at least 2 years naturally postmenopausal) must agree to utilize the same acceptable form of contraception from Screening through completion of the study.
* Subjects must be willing and able to comply with the study restrictions and requirements.
* Subjects or their parent or guardian must provide written informed consent and assent (where applicable) prior to participation in the study.

Exclusion Criteria:

* Patients enrolled in the previous Study RP103-03 who did not complete their last scheduled Study visit or who do not wish to continue on treatment with RP103.

AND for patients who did not complete the RP103-03 study:

* Subjects less than 1 year old
* Subjects with a known history, currently of the following conditions or other health issues that make it, in the opinion of the investigator, unsafe for them to participate: inflammatory bowel disease (if currently active) or have had prior resection of small intestine; Heart disease (e.g., myocardial infarction, heart failure, unstable arrhythmias or poorly controlled hypertension) 90 days prior to Screening; Active bleeding disorder 90 days prior to Screening; Malignant disease within the last 2 years.
* Patients with a hemoglobin level < 10 g/dL at Screening or a level that, in the opinion of the investigator, makes it unsafe for the subject to participate.
* Subjects with known hypersensitivity to cysteamine or penicillamine.
* Female subjects who are nursing, planning a pregnancy, known or suspected to be pregnant, or have a positive serum pregnancy screen.
* Subjects who, in the opinion of the Investigator, are not able or willing to comply with the protocol.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-08-27 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (10):
- United States (5):
  - California Pacific Medical Center (CPMC) Research Institute, San Francisco, California
  - Stanford University Medical School, Stanford, California
  - Emory Children's Center, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Texas Children's Hospital/Baylor University, Houston, Texas
- France (4):
  - Hospices Civils de Lyon, Lyon
  - Hôpital Arnaud Villeneuve - CHU Montpellier, Montpellier
  - Hopital Necker, Paris
  - Robert Debre Hospital, Paris
- Radboud University Nijmegen Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dohil R, Fidler M, Barshop BA, Gangoiti J, Deutsch R, Martin M, Schneider JA. Understanding intestinal cysteamine bitartrate absorption. J Pediatr. 2006 Jun;148(6):764-9. doi: 10.1016/j.jpeds.2006.01.050. PMID 16769383
- [Background] Fidler MC, Barshop BA, Gangoiti JA, Deutsch R, Martin M, Schneider JA, Dohil R. Pharmacokinetics of cysteamine bitartrate following gastrointestinal infusion. Br J Clin Pharmacol. 2007 Jan;63(1):36-40. doi: 10.1111/j.1365-2125.2006.02734.x. PMID 17229040
- [Background] Levtchenko EN, van Dael CM, de Graaf-Hess AC, Wilmer MJ, van den Heuvel LP, Monnens LA, Blom HJ. Strict cysteamine dose regimen is required to prevent nocturnal cystine accumulation in cystinosis. Pediatr Nephrol. 2006 Jan;21(1):110-3. doi: 10.1007/s00467-005-2052-0. Epub 2005 Oct 27. PMID 16252107
- [Derived] Langman CB, Greenbaum LA, Grimm P, Sarwal M, Niaudet P, Deschenes G, Cornelissen EA, Morin D, Cochat P, Elenberg E, Hanna C, Gaillard S, Bagger MJ, Rioux P. Quality of life is improved and kidney function preserved in patients with nephropathic cystinosis treated for 2 years with delayed-release cysteamine bitartrate. J Pediatr. 2014 Sep;165(3):528-33.e1. doi: 10.1016/j.jpeds.2014.05.013. Epub 2014 Jun 16. PMID 24948347
- See also: RP103 (marketed as PROCYSBI) is now approved by the US FDA for management of nephropathic cystinosis in patients 6 years and older. — http://procysbi.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initially, only patients who completed the previous Phase III Study RP103-03 (NCT01000961) were enrolled in this extension study. As of 27 September 2011, enrollment was opened up to additional participants, including children who were less than 6 years of age and kidney transplant subjects who qualified based on the inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | Cysteamine Bitartrate
Started | 60
Received Treatment | 59
Completed | 53
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (6.00)
Age, Customized [Count of Participants; unit: Participants]
  ≤ 6 years | 13
  > 6 to ≤ 12 years | 25
  > 12 to ≤ 21 years | 19
  > 21 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 58
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Drug-related adverse events (AEs) are AEs the investigator assessed as having relation to drug of 'possibly', 'probably' or 'definitely'.
  The severity of AEs was categorized according to the Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0 as follows:
  * Mild (Grade 1): experience is minor and does not cause significant discomfort to subject or change in activities of daily living (ADL); subject is aware of symptoms but symptoms are easily tolerated;
  * Moderate (Grade 2): experience is an inconvenience or concern to the subject and causes interference with ADL, but the subject is able to continue with ADL.
  * Severe (Grade 3): experience significantly interferes with ADL and the subject is incapacitated and/or unable to continue with ADL
  * Life-threatening (Grade 4): experience that, in the view of the Investigator, places the subject at immediate risk of death from the event as it occurred.
Time Frame: From first dose of study drug to 7 days after the last dose; median duration of treatment was 1461 days.
Population: All participants who received at least 1 dose of cysteamine bitartrate.
Measure: Count of Participants; unit: Participants
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 59
Participants
  Any adverse event | 58
  Adverse events related to study drug | 37
  Adverse events ≥ Grade 3 | 24
  Serious adverse events | 32
  Adverse events leading to discontinuation | 3

2. Secondary Outcome: Trough Plasma Cysteamine Concentration
Description: Plasma cysteamine concentration was determined using methods employing Hydrophilic Interaction Liquid Chromatography (HILC) high pressure liquid chromatography (HPLC) tandem mass spectrometry (HPLC-MS/MS).
Time Frame: Day 1 (predose) and Month 6, Years 1, 1.5, 2, 3, 4 and 5 at 0.5 hours post-dose
Population: The Pharmacokinetic/Pharmacodynamic (PK/PD) Population includes all participants who had at least one PK/PD measurement. Day 1 results only include participants who did not complete Study RP103-03.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 59
mg/L
  Day 1: number analyzed (Participants) | 19
  Day 1 | 0.17 (0.093)
  Month 6: number analyzed (Participants) | 56
  Month 6 | 0.29 (0.613)
  Year 1: number analyzed (Participants) | 56
  Year 1 | 0.37 (0.513)
  Year 1.5: number analyzed (Participants) | 55
  Year 1.5 | 0.48 (0.718)
  Year 2: number analyzed (Participants) | 45
  Year 2 | 0.36 (0.412)
  Year 3: number analyzed (Participants) | 28
  Year 3 | 0.34 (0.659)
  Year 4: number analyzed (Participants) | 38
  Year 4 | 0.47 (0.708)
  Year 5: number analyzed (Participants) | 26
  Year 5 | 0.40 (0.399)

3. Secondary Outcome: White Blood Cell Cystine Concentration
Description: White blood cell (WBC) cystine concentration was determined using high performance liquid chromatography-electrospray ionization tandem mass spectrometry (LC-ESI-MS/MS).
Time Frame: Day 1 (predose) and Month 6, Years 1, 1.5, 2, 3, 4 and 5 at 0.5 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol 1/2 Cystine/mg protein
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 59
nmol 1/2 Cystine/mg protein
  Day 1: number analyzed (Participants) | 18
  Day 1 | 1.68 (1.275)
  Month 6: number analyzed (Participants) | 56
  Month 6 | 0.93 (1.174)
  Year 1: number analyzed (Participants) | 55
  Year 1 | 0.65 (0.569)
  Year 1.5: number analyzed (Participants) | 54
  Year 1.5 | 0.75 (0.852)
  Year 2: number analyzed (Participants) | 44
  Year 2 | 0.65 (0.851)
  Year 3: number analyzed (Participants) | 28
  Year 3 | 0.66 (0.575)
  Year 4: number analyzed (Participants) | 28
  Year 4 | 1.38 (1.672)
  Year 5: number analyzed (Participants) | 24
  Year 5 | 1.17 (2.117)

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 7 days after last dose; median duration of treatment was 1461 days.
Arm/Group | Cysteamine Bitartrate
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 32/59
Other Adverse Events (participants affected / at risk) | 58/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cysteamine Bitartrate (N=59)
Appendicitis (Infections and infestations) | 7
Gastroenteritis (Infections and infestations) | 6
Appendicitis perforated (Infections and infestations) | 1
Bacterial diarrhoea (Infections and infestations) | 1
Otitis media chronic (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Salpingitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Urethritis (Infections and infestations) | 1
Renal failure chronic (Renal and urinary disorders) | 4
Renal failure (Renal and urinary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Renal tubular acidosis (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Gastric fistula (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 4
Acidosis (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 5
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 1
Biopsy kidney (Investigations) | 2
Investigation (Investigations) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Arnold-chiari malformation (Congenital, familial and genetic disorders) | 1
Cryptorchism (Congenital, familial and genetic disorders) | 1
Abnormal behavior (Psychiatric disorders) | 1
Impaired self-care (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Impaired healing (General disorders) | 1
Kidney transplant rejection (Immune system disorders) | 1
Convulsion (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Pseudoparalysis (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Nephrectomy (Surgical and medical procedures) | 1
Postoperative care (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cysteamine Bitartrate (N=59)
Vomiting (Gastrointestinal disorders) | 40
Diarrhoea (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 16
Abdominal pain (Gastrointestinal disorders) | 12
Breath odour (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 4
Abdominal discomfort (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Influenza (Infections and infestations) | 14
Nasopharyngitis (Infections and infestations) | 13
Gastroenteritis (Infections and infestations) | 11
Ear infection (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 10
Sinusitis (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 6
Bronchitis (Infections and infestations) | 5
Otitis media (Infections and infestations) | 5
Molluscum contagiosum (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 3
Pharyngitis streptococcal (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 3
Varicella (Infections and infestations) | 3
Viral infection (Infections and infestations) | 3
Headache (Nervous system disorders) | 22
Syncope (Nervous system disorders) | 5
Lethargy (Nervous system disorders) | 3
Fatigue (General disorders) | 10
Pyrexia (General disorders) | 8
Asthenia (General disorders) | 4
Influenza like illness (General disorders) | 4
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Joint sprain (Injury, poisoning and procedural complications) | 4
Arthropod bite (Injury, poisoning and procedural complications) | 3
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 6
Acne (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Conjunctivitis (Eye disorders) | 14
Photophobia (Eye disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 3
Blood creatinine increased (Investigations) | 5
Left ventricular hypertrophy (Cardiac disorders) | 4
Hypertension (Vascular disorders) | 7
Seasonal allergy (Immune system disorders) | 3
Depression (Psychiatric disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 4
Dysmenorrhoea (Reproductive system and breast disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT01197378/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT01197378/SAP_001.pdf